CLINICAL TRIAL: NCT06493747
Title: Efficacy and Mechanism Study of Acupuncture Combined With Neuromodulation Technology for Post-Stroke Aphasia Based on Multimodal Functional Magnetic Resonance Imaging
Brief Title: Acupuncture + Neuromodulation for Post-Stroke Aphasia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Yueyang Integrated Medicine Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-012
Record Dates: First submitted 2024-07-01; First posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Aphasia, Rehabilitation
MeSH Terms: conditions — Aphasia | interventions — Transcranial Magnetic Stimulation; Acupuncture Therapy; Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Combined Low- and High-Frequency rTMS Intervention (Experimental): Participants will receive a combined intervention of low-frequency rTMS (1Hz) and high-frequency rTMS (5Hz) using an 8-shaped coil, with each frequency's treatment duration and pulse count aligning with the protocol provided.
  Interventions: Device: Combined Low- and High-Frequency rTMS Intervention
- Combined High- and Low-Frequency rTMS Intervention (Experimental): Similar to Arm A, but the order of interventions is reversed, starting with high-frequency rTMS followed by low-frequency rTMS.
  Interventions: Device: Combined High- and Low-Frequency rTMS Intervention
- rTMS Experimental Group: Individualized Precision rTMS Therapy (Experimental): Participants will undergo individualized precision rTMS therapy based on integrated analysis of assessment data, with a continuous two-week intervention, 10-25 minutes per session, at an intensity of 80% of the active motor threshold (AMT).
  Interventions: Device: rTMS
- rTMS + Acupuncture Group: rTMS Combined with "Kaiqiao Jieyan" Acupuncture Therapy (Experimental): Participants will receive both the aforementioned rTMS therapy and "Kaiqiao Jieyan" acupuncture therapy, including specific acupoint selection and manipulation techniques.
  Interventions: Device: rTMS + Acupuncture
- rTMS Control Group: Conventional rTMS Intervention (Active Comparator): Participants will receive conventional rTMS intervention according to the guidelines' recommended strategies.
  Interventions: Device: rTMS
- Acupuncture Group: "Kaiqiao Jieyan" Acupuncture Therapy Alone (Active Comparator): Participants will receive only "Kaiqiao Jieyan" acupuncture therapy, without rTMS intervention.
  Interventions: Device: Acupuncture

INTERVENTIONS:
Device: Combined Low- and High-Frequency rTMS Intervention — This intervention involves the application of rTMS using an 8-shaped coil with a frequency of 1Hz for low-frequency stimulation and 5Hz for high-frequency stimulation, in accordance with the study protocol.
  Arms: Combined Low- and High-Frequency rTMS Intervention
Device: Combined High- and Low-Frequency rTMS Intervention — Similar to Arm A, but the sequence of low and high-frequency rTMS is reversed.
  Arms: Combined High- and Low-Frequency rTMS Intervention
Device: rTMS — Participants receive an individualized rTMS therapy plan based on integrated analysis of assessment data, targeting specific brain areas to enhance language function recovery post-stroke.
  Arms: rTMS Experimental Group: Individualized Precision rTMS Therapy
Device: rTMS + Acupuncture — Participants undergo a combined treatment of rTMS as described for the rTMS Experimental Group and traditional Chinese acupuncture based on the "Kaiqiao Jieyan" method, targeting specific acupoints to facilitate recovery.
  Arms: rTMS + Acupuncture Group: rTMS Combined with "Kaiqiao Jieyan" Acupuncture Therapy
Device: rTMS — Participants receive a conventional rTMS treatment as per established guidelines, serving as an active comparator to the experimental interventions.
  Other Names: Control Group
  Arms: rTMS Control Group: Conventional rTMS Intervention
Device: Acupuncture — Participants receive "Kaiqiao Jieyan" acupuncture therapy alone, without rTMS, following traditional Chinese medicine protocols for post-stroke aphasia rehabilitation.
  Arms: Acupuncture Group: "Kaiqiao Jieyan" Acupuncture Therapy Alone

SUMMARY:
The aim of this clinical trial is to assess the therapeutic efficacy of acupuncture combined with neuromodulation techniques for the treatment of post-stroke aphasia and to explore the brain mechanisms involved. The study seeks to answer two primary questions: the effectiveness of the integrated intervention of acupuncture and repetitive transcranial magnetic stimulation (rTMS) on post-stroke aphasia, and the mechanisms underlying language function impairment and recovery.

The research is divided into two parts:

Part One:

Participants will be randomized into two groups:

Group A: Receives low-frequency rTMS followed by high-frequency rTMS. Group B: Receives high-frequency rTMS followed by low-frequency rTMS.

Part Two:

Participants will be randomized into four groups:

rTMS Experimental Group: Individualized targets and intervention methods based on integrated fMRI and behavioral data. The rTMS intervention involves continuous treatment for two weeks, 5 sessions per week, each lasting 10-25 minutes, at 80% of the active motor threshold (AMT).

rTMS Control Group: Standard rTMS protocol guided by clinical recommendations, with continuous treatment for two weeks, 5 sessions per week, each 20 minutes, at 80% AMT.

Electroacupuncture Group: Points include Speech Area 1 (Yan Yu Yi Qu 1), Speech Area 2 (Yan Yu Yi Qu 2), Fengchi (Fengchi, GB20), Tiantu (Tiantu, CV22), Tongli (Tongli, HT5), Lianquan (Lianquan, CV23), and Paralianquan (Pang Lianquan). After needle insertion and obtaining Qi, electrical stimulation is applied with a discontinuous wave at 2Hz, at a tolerable intensity for the patient, for 30 minutes each session.

Combined rTMS and Electroacupuncture Group: Combines both intervention methods as described above.

DETAILED DESCRIPTION:
Aphasia is a severe disabling consequence of stroke, typically caused by damage to the cortical and subcortical structures perfused by the left middle cerebral artery. Studies have indicated that over 20% of stroke patients develop aphasia. Although most patients exhibit some degree of spontaneous recovery within the first month after stroke, a significant number still suffer from chronic deficits six months post-stroke. Conventional rehabilitation methods and traditional Chinese medicine techniques often encounter efficacy plateaus in the treatment process. Therefore, there is an urgent need for innovative language therapy strategies to maximize recovery from aphasia. Non-invasive brain stimulation techniques, such as transcranial magnetic stimulation (TMS), have the potential to modulate cortical excitability and plasticity. Acupuncture therapy can activate language neural functions, establish collateral cerebral vascular circulation, and reconstruct the neural circuitry of language motor control. However, when facing patients with complex post-stroke aphasia, there are certain limitations. This study employs a randomized, blinded, controlled clinical design to verify the therapeutic efficacy of acupuncture combined with transcranial magnetic stimulation in treating post-stroke aphasia and to explore the underlying brain mechanisms of recovery.

The research is divided into two parts:

Part One:

Participants will be randomized into two groups:

Group A: Receives low-frequency rTMS followed by high-frequency rTMS. Group B: Receives high-frequency rTMS followed by low-frequency rTMS.

Part Two:

Participants will be randomized into four groups:

rTMS Experimental Group: Individualized targets and intervention methods based on integrated fMRI and behavioral data. The rTMS intervention involves continuous treatment for two weeks, 5 sessions per week, each lasting 10-25 minutes, at 80% of the active motor threshold (AMT).

rTMS Control Group: Standard rTMS protocol guided by clinical recommendations, with continuous treatment for two weeks, 5 sessions per week, each 20 minutes, at 80% AMT.

Electroacupuncture Group: Points include Speech Area 1 (Yan Yu Yi Qu 1), Speech Area 2 (Yan Yu Yi Qu 2), Fengchi (Fengchi, GB20), Tiantu (Tiantu, CV22), Tongli (Tongli, HT5), Lianquan (Lianquan, CV23), and Paralianquan (Pang Lianquan). After needle insertion and obtaining Qi, electrical stimulation is applied with a discontinuous wave at 2Hz, at a tolerable intensity for the patient, for 30 minutes each session.

Combined rTMS and Electroacupuncture Group: Combines both intervention methods as described above.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with aphasia following stroke according to both traditional Chinese and Western medical standards; first-time stroke in the left cerebral hemisphere (including cerebral infarction and cerebral hemorrhage), with unilateral lesion.
2. Age between 25 and 75 years old, disease course of at least 1 month, no gender restrictions.
3. Right-handed as tested by the Edinburgh Handness Inventory, with at least an elementary school education level.
4. Retention of basic cognitive functions such as attention, memory, and visuospatial skills (Non-language-based Cognitive Assessment, NLCA score >70).
5. Aphasia confirmed by initial assessment with the Western Aphasia Battery (WAB); an Aphasia Quotient (AQ) <93.8 indicates aphasia.
6. Possess a certain level of auditory comprehension and can tolerate research examinations lasting 0.5-1 hour.
7. The subject and their legal guardian understand and consent to participate in this study and have jointly signed the informed consent form.

Exclusion Criteria:

1. Moderate to severe dysarthria as assessed by the Frenchay Dysarthria Assessment.
2. Severe speech apraxia or oral-facial apraxia.
3. Significant anxiety or moderate to severe depressive symptoms as assessed by the Hamilton Anxiety and Depression Scales.
4. Pre-stroke speech or language disorders.
5. Severe systemic diseases such as cardiopulmonary diseases that cannot tolerate rehabilitation treatment or infectious diseases.
6. Significant sleep disorders or mental disorders.
7. Pregnant or lactating women.
8. Contraindications for MRI examination (presence of metal foreign bodies or other implanted electronic devices in the body).

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Western Aphasia Battery (WAB) | Baseline: Pre-intervention assessment. Immediately Post-Intervention: Assessment at the end of the 2-week intervention. Follow-Up Assessments: Assessments are also conducted at 1, 2, and 3 months post-intervention.
  Western Aphasia Battery (WAB): Assesses aphasia severity in speech, comprehension, reading, and writing. Score Range: WAB-derived AQ scores range from 0 (severe impairment) to 100 (no impairment). Interpretation: Higher AQ scores on the WAB indicate better language function in aphasia patients.

SECONDARY OUTCOMES:
Token Test (Abbreviated Version) | Baseline: Pre-intervention assessment. Immediately Post-Intervention: Assessment at the end of the 2-week intervention. Follow-Up Assessments: Assessments are also conducted at 1, 2, and 3 months post-intervention.
  Token Test (Abbreviated Version): The abbreviated Token Test will be utilized to evaluate patients' spoken language comprehension and abstract thinking abilities. This assessment will provide insights into the participants' cognitive and linguistic capacities.
Boston Naming Test | Baseline: Pre-intervention assessment. Immediately Post-Intervention: Assessment at the end of the 2-week intervention. Follow-Up Assessments: Assessments are also conducted at 1, 2, and 3 months post-intervention.
  The Boston Naming Test will evaluate patients' ability to name 30 common items from pictures, measuring improvements in naming abilities.
American Speech-Language-Hearing Association Functional Assessment of Communication Skills for Adults (ASHA FACS). | Baseline: Pre-intervention assessment. Immediately Post-Intervention: Assessment at the end of the 2-week intervention. Follow-Up Assessments: Assessments are also conducted at 1, 2, and 3 months post-intervention.
  ASHA FACS assesses functional communication in aphasia, including basic needs and social integration. Score Range - Communicative Independence Scale: 1 (maximal assistance) to 7 (independence) across 43 items. Score Range - Qualitative Dimensions Scale: 1 (poor quality) to 5 (excellent quality). Interpretation: Higher scores indicate better communication outcomes in aphasia.
Stroke-Specific Quality of Life Scale (SS-QOL) | Baseline: Pre-intervention assessment. Immediately Post-Intervention: Assessment at the end of the 2-week intervention. Follow-Up Assessments: Assessments are also conducted at 1, 2, and 3 months post-intervention.
  The Stroke-Specific Quality of Life Scale (SS-QOL) is used to evaluate the health-related quality of life in stroke patients, focusing on the specific impacts of stroke on daily living and well-being. Scale Title: Stroke-Specific Quality of Life Scale (SS-QOL). Score Range: The SS-QOL score ranges from 1.0 (lowest quality of life) to 5.0 (highest quality of life). Interpretation: Higher scores indicate a better quality of life for stroke survivors.
Multimodal MRI Assessment | Baseline: Pre-intervention assessment. Immediately Post-Intervention: Assessment at the end of the 2-week intervention. Follow-Up Assessments: Assessments are also conducted at 1, 2, and 3 months post-intervention.
  This includes 3D structural MRI (sMRI), functional MRI (fMRI) during task performance and at rest, and Diffusion Tensor Imaging (DTI) to evaluate changes in brain structure and function.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Yueyang Integrated Medicine Hospital, Shanghai, Shanghai Municipality, China